CLINICAL TRIAL: NCT00022971
Title: Combination Antibody Therapy With Apolizumab (1D10) and Rituximab (CD20) in Relapsed Lymphoma and CLL
Brief Title: Combination Antibody Therapy for Relapsed Lymphoma and Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010235; 01-C-0235; NCT00029367 (obsolete NCT alias)
Record Dates: First submitted 2001-08-17; First posted 2001-08-20 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2017-03-17

CONDITIONS: Diffuse Large B-Cell Lymphoma; Follicular Lymphoma; Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma; Small Lymphocytic Lymphoma
Keywords: Monoclonal Antibody; Lymphoma; Rituximab; Hu1D10; Non-Hodgkin's Lymphoma; NHL; Chronic Lymphocytic Leukemia; CLL; Leukemia
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma; Lymphoma, Non-Hodgkin; Leukemia | interventions — apolizumab; Rituximab

ARMS (1):
- 1 (Experimental): Apolizumab followed by rituixmab every 4 weeks
  Interventions: Biological: Apolizumab; Biological: Rituximab

INTERVENTIONS:
Biological: Apolizumab — Apolizumab IV on Day 1. Administer weekly for 4 weeks
Biological: Rituximab — Rituximab IV 24-36 hours after Apolizumab ends. Administer weekly for 4 weeks

SUMMARY:
This study will evaluate the safety and effectiveness of a combination of two antibodies, apolizumab and rituximab (Rituxan ), in treating B-cell lymphomas and chronic lymphocytic leukemia. Rituximab attaches to a molecule called CD20 on B-cell lymphomas and can cause significant shrinkage of these tumors in up to half of patients. However, it does not cure the lymphoma, which usually returns. Also, it is not as effective against leukemia. Apolizumab attaches to a protein called 1D10 on B-cell cancers and has also been able to shrink tumors in some patients. There is little experience apolizumab in patients with leukemia. This study will test whether the two antibodies together are more effective against these tumors than either one alone.

Patients 18 years and older with B-cell lymphoma or chronic lymphocytic leukemia may be eligible for this study. Patients' leukemia or lymphoma cells must have both the CD20 and 1D10 antigen receptors and must have had at least one systemic treatment for their disease. Candidates are screened with a medical history and physical examination, blood and urine tests, electrocardiogram, x-rays and other imaging studies, and possibly a bone marrow aspirate (withdrawal of a small marrow sample through a needle inserted into the hip bone) and lumbar puncture (withdrawal of a small sample of cerebrospinal fluid-fluid that bathes the brain and spinal cord-through a needle placed between the bones in the lower back).

Participants receive infusions of rituximab and apolizumab once a week for 4 weeks. The first patients in the study receive lower doses of apolizumab with standard doses of rituximab. If the apolizumab is well tolerated, subsequent patients are given higher doses. Patients are also given dexamethasone or another similar steroid, diphenhydramine (Benadryl ), and acetominophen (Tylenol ) to reduce reactions to the antibodies. After 4 weeks of treatment, patients are followed frequently to examine the response to treatment and evaluate drug side effects. Patients whose tumors do not grow during the 4 weeks of therapy may be offered another course of treatment at a later time. Participants are followed periodically after treatment ends until their disease worsens or the study ends.

...

DETAILED DESCRIPTION:
While recurrent non-Hodgkin's lymphoma (NHL) and chronic lymphocytic leukemia (CLL) are often responsive to therapy, they are rarely curable and disease control is the primary therapeutic goal. Rituximab, a chimeric anti-CD20 monoclonal antibody, has shown single agent activity in these diseases and is currently approved for the therapy of recurrent indolent lymphoma. However, rituximab induces objective remission in at most 60% of cases with inevitable relapse. The 1D10 antigen, a subclass of the HLA-DR molecule, is expressed in a majority of cases of B-cell malignancy. Apolizumab is a humanized monoclonal antibody that targets this antigen. In a phase I dose escalation trial this antibody has shown clinical activity against B-cell NHL that express the 1D10 antigen. Acute infusional toxicity has been tolerable, and a maximum of 5 mg/kg has been given in each of 4 weekly doses. Preclinical in vitro data from Dr. George Weiner's laboratory suggests at least additive anti-tumor efficacy when cells are exposed to both antibodies simultaneously. This trial will pilot the use of combination therapy with rituximab and apolizumab in patients with tumors that express both antigens. Feasibility and tolerability of the regimen will be determined. Experimental endpoints will include pharmacokinetics of apolizumab, assessment of apoptosis in circulating CLL cells by FACS analysis with Annexin 5, assessment of T-and B-cell dynamics, and effects of rituximab and apolizumab on CLL mRNA as measured by cDNA microarray. Following the first 21 patients on trial, the administration sequence of rituximab and apolizumab was changed from rituximab first to apolizumab first to potentially reduce sensitization of apolizumab toxicity by rituximab.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of B-cell lymphoma, Waldenstrom's CLL with surface expression of both CD20 and 1D10 antigen by immunohistochemistry (IHC) or fluorescence of activated cell sorting (FACS) with anti-CD20 and 1D10 antibody. Positive 1D10 expression in a FACS assay is defined as more than 2 times the mean fluorescence intensity (MFI) of the control antibody by FACS or greater than 20% of cells 1D10+ by IHC.

Confirmation of diagnosis in Laboratory of Pathology, NCI or OSU.

Prior therapy with at least one systemic treatment, and not a candidate for potentially curative (i.e., transplant) treatment at the time of study entry. Prior treatment with rituximab greater than or equal to 1 month ago is permitted.

Age greater than 18 years.

ECOG performance status less than or equal to 2.

Major organ function: ANC greater than or equal to 500/microliter, Platelet greater than or equal 25,000/microliter, Creatinine less than or equal to 1.5 mg/dl or creatinine clearance greater than 60 cc/min; SGPT less than 5 x upper limit of normal; bilirubin less than 2 mg/dl (total) except less than 5 mg/dl in patients with Gilbert's syndrome as defined by greater than 80% unconjugated; unless impairment due to organ involvement by lymphoma.

Provides informed consent.

EXCLUSION CRITERIA:

Pregnancy or nursing. Both male and female patients must be willing to use adequate contraception.

Prior apolizumab treatment.

SActive cardiac disease, cerebrovascular disease or peripheral arterial vascular disease.

Active CNS lymphoma.

Systemic cytotoxic chemotherapy within 3 weeks of enrollment or systemic steroids (except stable doses less than 10 mg/day) within 1 week of enrollment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-08-15; Primary Completion 2010-01-22 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
MTD | After one cycle

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H Wilson, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Shan D, Ledbetter JA, Press OW. Apoptosis of malignant human B cells by ligation of CD20 with monoclonal antibodies. Blood. 1998 Mar 1;91(5):1644-52. PMID 9473230
- [Background] McLaughlin P. Inroads in the therapy of indolent lymphomas: exploiting biological insights. Cancer Invest. 1999;17(1):73-86. No abstract available. PMID 10999051
- [Background] Weiner LM. Monoclonal antibody therapy of cancer. Semin Oncol. 1999 Oct;26(5 Suppl 14):43-51. PMID 10561017